CLINICAL TRIAL: NCT04423068
Title: Intervention to Facilitate Contraception Provision by Pediatric Hospitalists: A Feasibility Study
Brief Title: Inpatient Adolescent Contraception
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Children's Mercy Hospital Kansas City (Other)
Responsible Party: Principal Investigator, Abbey Masonbrink, Physician, Hospital Medicine, Children's Mercy Hospital Kansas City
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00001115
Record Dates: First submitted 2020-06-05; First posted 2020-06-09 (Actual); Last update posted 2023-04-05 (Actual); Status verified 2023-04

CONDITIONS: Pregnancy Related; Contraception; Contraceptive Usage; Contraception Behavior; Pregnancy
Keywords: LARC; Long acting reversible contraception
MeSH Terms: conditions — Contraception Behavior | interventions — Contraceptive Agents

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Overall Study (Experimental)
  Interventions: Behavioral: SexHealth II; Drug: Contraceptive

INTERVENTIONS:
Behavioral: SexHealth II — SexHealth II is an intervention that will focus exclusively on provision of hormonal contraception counseling and provision for hospitalized female adolescents
Drug: Contraceptive — The investigators will offer initiation of the following contraceptives:
  Ethinyl Estradiol and Etonogestrel 0.015mg-0.12mg vaginal ring (Nuva Ring) Etonogestrel 68mg subcutaneous implant (Nexplanon) Medroxyprogesterone 150mg/ml 150 mg IM injection Ethinyl Estradiol and Norgestimate (Sprintec) 35mcg-0.25mg tablet Norelgestromin/Ethinyl estradiol transdermal patch (Ortho Evra) Norethindrone 0.35mg tablet
  Emergency Contraception:
  Ulipristal 30 mg tablet Levonorgestrel 1.5mg tablet

SUMMARY:
The overall goal of this study is to refine and pilot test the investigators novel intervention to offer contraception counseling and initiation for hospitalized female adolescents, focusing on long acting reversible contraception (LARC).

DETAILED DESCRIPTION:
There are two primary objectives in this study. The first objective is to refine the investigators previously developed general sexual risk reduction intervention (SexHealth II) to focus on patient-centered contraception counseling and initiation for hospitalized female adolescents. The second objective is to conduct an open trial to assess feasibility of the investigators SexHealth II intervention among hospitalized females aged 14-21 years (N=75). Among key stakeholders (i.e., adolescent participants, parents/guardians, hospitalists and nurses), the investigators will assess Bowen's feasibility constructs: acceptability, demand, implementation, practicality, integration, and limited-efficacy testing. The investigators hypothesize that the SexHealth II intervention will be deemed feasible by female adolescent participants (i.e., the median score across all feasibility items will be > 2.5.)

ELIGIBILITY:
Inclusion Criteria:

* Adolescents who are biologically female and have reproductive potential (14-21 years old) admitted to the general pediatric hospitalist service will be eligible.
* A convenience sample of parents/guardians of enrolled participants who are English speaking will be eligible for post-intervention feasibility survey. Parent consent or enrollment in the study is not required for female adolescent enrollment.
* A convenience sample of hospitalists and nurses caring for enrolled participants and the health educator will be eligible for the post-intervention feasibility study.

Exclusion Criteria:

* Subjects who are determined to be too ill, have severe psychiatric illness or cognitive impairment (based on hospitalist assessment), are seeking care related to sexual assault, or are not able to speak English fluently will not be eligible.
* Parents/guardians, hospitalists, health educator and nurses who are not able to speak English fluently will not be eligible for post-intervention feasibility survey.

  * Adults unable to consent - Exclude
  * Individuals who are not yet adults (infants, children, teenagers) - Include
  * Pregnant women - Exclude
  * Prisoners - Exclude
  * Wards of the state - Include

Withdraw Criteria:

- Subjects who are screened and report no sexual activity (past or anticipated "unlikely"/"very likely" within few weeks to months) will be withdrawn from the study.

Ages: 14 Years to 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 25 (Actual)
Dates: Start 2020-12-10 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2023-04-04 (Actual)

PRIMARY OUTCOMES:
Feasibility of SexHealth II, an intervention to provide contraception counseling and initiation among hospitalized female adolescents | 3 months
  The investigators primary outcome is feasibility of the intervention among female adolescent participants, which the investigators will assess by administering a survey with 12 Likert-type items with responses ranging from 0 (strongly disagree) to 4 (strongly agree). The midpoint (neutral) point on the 0-4 scale is 2, and the investigators define "acceptable level of feasibility" as the median feasibility rating in the population exceeding 2.5, meaning at least half the ratings are positive. Thus, the investigators will test the hypothesis that the true median feasibility rating in the population of adolescents from which the sample is drawn is greater than 2.5.
  The investigators expect the true median is above 2.5. Assuming its value is conservatively 2.75, a sample size of 75 provides 90% power to reject H0 using a two-sided sign test for the population median.

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Mercy Hospitals and Clinics, Kansas City, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Masonbrink AR, Noel-MacDonnell J, Staggs VS, Stancil S, Goggin K, Miller MK. Feasibility of a Contraception Intervention for Hospitalized Adolescents and Young Adults. Hosp Pediatr. 2023 Apr 1;13(4):337-344. doi: 10.1542/hpeds.2022-006996. PMID 36897226